CLINICAL TRIAL: NCT06261736
Title: The Effectiveness of Prophylactic Antibiotics for Urethral Bulking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Erika Wasenda, MD, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2107044-1
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Stress Urinary Incontinence; Postoperative Urinary Tract Infection; Urethral Bulking
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic Group (Experimental): Those randomized to this group will receive a one-time dose of an oral antibiotic prior to the urethral bulking procedure. The antibiotic will be based on the participants' allergies, medical history, and current medication list.
  Interventions: Other: Prophylactic antibiotics
- No antibiotic group (Other): Those randomized to this group will not receive an antibiotic prior to the urethral bulking procedure.
  Interventions: Other: No antibiotics

INTERVENTIONS:
Other: Prophylactic antibiotics — These participants will be given a single dose of an oral antibiotic prior to the procedure.
  Arms: Antibiotic Group
Other: No antibiotics — These participants will not be given an antibiotic prior to the procedure.
  Arms: No antibiotic group

SUMMARY:
The goal of this clinical trial is to evaluate if prophylactic antibiotics in urethral bulking are effective in reducing postprocedural urinary tract infections.

DETAILED DESCRIPTION:
Urethral bulking is a minimally invasive surgical treatment option for stress urinary incontinence (SUI). One commonly reported post-procedural complication is urinary tract infection (UTI). UTI rates are variable where studies have reported rates from as low as 0% to as high as 40%. Along with this variability, the instructional inserts for various bulking agents have inconsistent recommendations for use of prophylactic antibiotics. The American Urologic Association recommends antimicrobial prophylaxis for cystourethroscopy procedures involving minor manipulation. Currently, there are no clear guidelines regarding the utility of prophylactic antibiotics for urethral bulking. The objective of our study is to determine the effectiveness of prophylactic antibiotics in urethral bulking for reducing post procedural UTIs.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo a urethral bulking procedure
* Age 18 ≥ over

Exclusion Criteria:

* History of recurrent urinary tract infections
* Known history of urinary retention
* Allergies or contraindications to multiple antibiotics
* Inability to tolerate oral antibiotics
* Concomitant surgical procedures at the time of urethral bulking
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of urinary tract infection (UTI) | Within 4 weeks after the procedure
  The rate of UTI based on symptoms and a positive urine culture

SECONDARY OUTCOMES:
Rate of postoperative urinary retention | Within 4 weeks after the procedure
  The rate of postoperative urinary retention
Rates of other postoperative complications | Within 4 weeks after the procedure
  The rate of other complications (bleeding, discomfort, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Wasenda, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Health, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No